CLINICAL TRIAL: NCT00863551
Title: Sanctura Muscarinic Receptor Antagonist Resists Transport (SMART) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-SXR-09-001; SMART Trial (Other: Allergan)
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Elderly; Pharmacokinetics; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — trospium chloride

ARMS (1):
- Trospium Chloride Extended Release, 60 mg (Experimental): Trospium Chloride Extended Release, 60 mg
  Interventions: Drug: Trospium Chloride

INTERVENTIONS:
Drug: Trospium Chloride — Extended release, 60 mg, oral daily
  Other Names: Sanctura XR™ 60 mg

SUMMARY:
This study evaluates the penetration through the blood-brain-barrier of trospium chloride at plasma steady state (Day 10) in elderly subjects with overactive bladder symptoms. Trospium levels in cerebrospinal fluid (CSF) and peak and trough plasma levels will be measured. Baseline and day 10 post-dose neurocognitive testing will be compared using a reliable change index to assess if any study subject shows evidence of a clinically and statistically significant change in memory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 65-75 years of age without evidence of memory impairment
* Subject has overactive bladder symptoms but otherwise healthy
* Non-smoker (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the screening visit)
* Weight within normal range
* Ability to follow study instructions and likely to complete all required visits

Exclusion Criteria:

* Residual urine within bladder greater than 4 ounces
* Moderate or severe memory impairment
* Bleeding disorder
* Blood-thinning agents
* Concurrent overactive bladder medication
* Concurrent dementia drugs: Aricept (donepezil), Namenda (memantine), Cognex (tacrine), Exelon (rivastigmine), Razadyne (galantamine), galantamine or similar drugs for dementia
* Chronic kidney failure
* Abdominal bypass surgery for obesity

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trospium Chloride Extended Release, 60 mg
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trospium Chloride Extended Release, 60 mg
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 68 [65 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Spinal Fluid Levels of Trospium at Day 10, Hour 5
Description: Cerebral spinal fluid levels of Trospium at day 10, hour 5. Cerebral spinal fluid was collected from each patient.
Time Frame: Day 10, Hour 5
Population: Intent-to-treat, which included all patients who started the study.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Trospium Chloride Extended Release, 60 mg
Number analyzed (Participants) | 12
Picograms per milliliter (pg/mL) | NA (NA) — The data were below the limit of quantitation (BLQ).

2. Secondary Outcome: Percentage of Study Subjects With No Clinically Significant Effect on Neurocognitive Function Total Recall Score as Measured by the Hopkins Verbal Learning Test-Revised (HVLT-R) at Day 10 Post-Dose
Description: The HVLT-R is an instrument used to measure verbal learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and yes/no delayed recognition. The total recall score was the sum of 3 'free recall' learning trials, and reflects the patient's ability to learn. The total score ranges from 0 (no memory) to 36 (best memory).
Time Frame: Day 10
Population: Intent-to-treat, which included all patients who started the study.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Trospium Chloride Extended Release, 60 mg
Number analyzed (Participants) | 12
Percentage of Subjects | 100

3. Secondary Outcome: Percentage of Study Subjects With No Clinically Significant Effect on Neurocognitive Function Delayed Recall Score as Measured by the Hopkins Verbal Learning Test-Revised (HVLT-R) at Day 10 Post-Dose
Description: The HVLT-R is an instrument used to measure verbal learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and yes/no delayed recognition trial. The delayed recall score provides a measure of the patient's recent memory. The total score ranges from 0 (no memory) to 12 (best memory).
Time Frame: Day 10
Population: Intent-to-treat, which included all patients who started the study.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Trospium Chloride Extended Release, 60 mg
Number analyzed (Participants) | 12
Percentage of Subjects | 91.7

4. Secondary Outcome: Percentage of Study Subjects With No Clinically Significant Effect on Neurocognitive Function as Measured by the Brief Visuospatial Memory Test-Revised (BVMT-R) Total Score at Day 10 Post-Dose
Description: The BVMT-R is an instrument used to measure visual learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and yes/no delayed recognition trial. The total recall score is the sum of 3 free recall learning trials, and reflects the patient's ability to learn. The total score ranges from 0 (no memory) to 12 (best memory). Due to technical problems associated with the administration of the test, the results were invalid.
Time Frame: Day 10
Population: Intent-to-treat, which included all patients who started the study. Due to technical problems associated with the administration of the test, the results were invalid.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Trospium Chloride Extended Release, 60 mg
Number analyzed (Participants) | 12
Percentage of Subjects | NA — Due to technical problems associated with the administration of the test, the results were invalid.

5. Secondary Outcome: Percentage of Study Subjects With No Clinically Significant Effect on Neurocognitive Function as Measured by the Brief Visuospatial Memory Test-Revised (BVMT-R) Delayed Recall Score at Day 10 Post-Dose
Description: The BVMT-R is an instrument used to measure visual learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and a yes/no delayed recognition trial. The delayed recall score, derived from the delayed recall trial, provides a measure of the patient's recent memory. The total score ranges from 0 (no memory) to 12 (best memory). Due to technical problems associated with the administration of the test, the results were invalid.
Time Frame: Day 10
Population: as for outcome 4
Measure: Number; unit: Percentage of Subjects
Arm/Group | Trospium Chloride Extended Release, 60 mg
Number analyzed (Participants) | 12
Percentage of Subjects | NA — Due to technical problems associated with the administration of the test, the results were invalid.

ADVERSE EVENTS:
Arm/Group | Trospium Chloride Extended Release, 60 mg
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trospium Chloride Extended Release, 60 mg (N=12)
Headache (Nervous system disorders) | 7
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Low back pain (Musculoskeletal and connective tissue disorders) | 2
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Change in taste (General disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
Due to technical problems associated with the administration of the BVMT-R test, the results were invalid, therefore, results for Outcome Measures 4 and 5 are not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo